CLINICAL TRIAL: NCT03053791
Title: A Phase I/II Open-label Multicenter Trial to Evaluate Safety and Preliminary Efficacy of Unilateral Deep Brain Stimulation of the Mesencephalic Locomotor Region in Patients With Incomplete Spinal Cord Injury
Brief Title: Deep Brain Stimulation in Patients With Incomplete Spinal Cord Injury for Improvement of Gait
Acronym: DBS-SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Balgrist University Hospital (Other); ETH Zurich (Other); Wings for Life (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNCTP000000598
Record Dates: First submitted 2016-04-26; First posted 2017-02-15 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injury
Keywords: Deep brain stimulation; DBS; Spinal cord injury; SCI; Paraplegia; Mesencephalic locomotor region; MLR; Pedunculopontine nucleus; PPN
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Single group of patients with spinal cord injury and spared fibers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Single-armed study. All patients will receive treatment.
  Interventions: Procedure: Deep brain stimulation in mesencephalic locomotor region; Device: Implantation of a Deep brain stimulation system

INTERVENTIONS:
Procedure: Deep brain stimulation in mesencephalic locomotor region — Implantation of Electrodes in the Mesencephalic Locomotor Region for improvement of Locomotion and Gait
Device: Implantation of a Deep brain stimulation system — Implantation of a Medtronic Percept PC Impulse Generator for chronic Stimulation of the selected target.

SUMMARY:
Spinal cord injuries are anatomically mostly incomplete, showing tissue bridges of the spinal cord at the injury site. Of the 60% functionally incomplete patients, about half face a life in the wheelchair. Besides conventional rehabilitation, no prominsing further treatment options exist. One of the most plastic systems involved in locomotion is the pontomedullary reticulospinal tract, which is the oldest locomotor command system existing in most vertebrates, including primates. Muscle activation patterns for limb movements are programmed in the spinal cord and have to be activated and coordinated through commands from the so called mesencephalic locomotor region (MLR). The MLR consists of nerve cells in the lower mesencephalic tegmentum sending uni- and bilateral signals through the medullary reticulospinal tracts. Classical physiological studies showed that electrical stimulation of the MLR induce locomotion. For the first time this approach was transferred and recently published in a model of induced incomplete spinal cord injury by the Schwab group. Rats severly impaired in motor hindlimb control with only 10-20% spared white matter, recovered with fully functional weight bearing locomotion under MLR deep brain stimulation (DBS). Even rats with only 2-10% spared white matter regained weight supporting stepping. DBS is a clinical standard treatment option in patients with movement disorders but does not relieve all symptoms. Therefore, small studies of MLR stimulations have been safely used in Parkinsonian patients showing freezing of gait and frequent falls with variable results. In a translational approach, we aim at performing a multidisciplinary phase one clinical trial with 5 patients and incomplete spinal cord injury. With the means of our established universitary setup for DBS treatments the operations will be performed unilaterally under local anaesthesia in the Division of Neurosurgery, USZ, with perioperative electrophysiological recordings, clinical assessments and gait analysis under test stimulation in the Spinal Cord Injury Center Balgrist.

DETAILED DESCRIPTION:
After approval by the local ethics committee we will perform a phase I open-label trial to evaluate safety and preliminary efficacy of unilateral deep brain stimulation of the mesencephalic locomotor region in patients with incomplete spinal cord injury. Male or female subjects (18-75 year-old) with completed in-patient rehabilitation will be enrolled for screening evaluations at minimum 3 months post-injury. DBS operation will be performed at minimum 3 months post-injury. Primary endpoint will be improvement of locomotion as determined by the 6-Minute walking test.

Secondary endpoints will be electrophysiological/clinical and image based characterization of the mesencephalic locomotor region, questionnaire based/ professional assessments of quality of life, pain, micturition, sleep behavior, cognitive function and psychiatric evaluations (mood, anxiety, impulse control, delusional and affective disorders). The study population will consist of 5 subjects and the study period for each patient is 6 months postoperatively. Briefly, candidate subjects, able to stand with a walker or 2 crutches and with stable neurological condition will have to meet all of the inclusion and none of the exclusion criteria. Subjects will have preoperative examinations (e.g. MRI scans of the head and spine, neuropsychological, psychiatric and sleep status etc.) according to our standard protocols of DBS for movement disorders, especially Parkinson's disease, based on certification criteria of Highly-Specialized-Medicine DBS centers in Switzerland. Neurological assessments for spinal cord injury impairment as defined by study protocol will be performed at the University Hospital Balgrist.

The operation will be performed in the Division of Neurosurgeon by the neurosurgical PI of this study: awake subjects will have their heads fixed in a stereotactic ring with local anesthesia and high resolution head scans will be performed to define the stereotactic space for targeting through anatomical landmarks defined on individual MRI as described in the literature. In contrast to bilateral implantations in Parkinsonian patients, here, a single burr hole will be opened under local anesthesia on the contralateral side of the worse lower extremity of the subject. Microelectrode recordings of single-cells as well as local field potentials will be mapped starting 1 cm prior the MLR target. Four states will be analyzed: resting state, imagination of walking, passive and active lower limb movement. These recordings will help to further determine the places of stimulation as the next step of surgery. Here, slow increases of the stimulation amplitude with a constant frequency of e.g. 50Hz will be applied to determine activation of lower limb muscle activity with electroneuromyographic recordings and detection of possible amelioration of intended active movements. Since the subject is awake, possible side effects will be professionally monitored at each site of stimulation and amplitude. Next, the electrode for recording and stimulation will be exchanged with the standard 8-contact directional DBS electrode for Parkinson's disease patients (1.28 mm in diameter, 1.5mm length of each contact and 0.5 mm spacing in between). All subjects will receive an intraoperative head scan to verify correct placement and accuracy. If refinement is not necessary, the first operative procedure will be regarded as finished and the subject will be transferred to the intermediate care unit overnight to recover from surgery. The surgeon will decide, if the impulse generator will be implanted in the same surgery or delayed. Subjects will undergo regular assessments until discharge and further on in an outpatient setup around day 30 post-surgery, as well as 3 and 6 months afterwards. Rehabilitative postoperative treatment will be assisted by using the recently CE certificated and award winning FLOAT system ("Free Levitation for Overground Active Training") which allows robotic multidirectional relief of body weight and exact gait/posture analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent
2. Participation in two assessment sessions before enrollment (Screening and baseline)
3. Willingness and ability to comply with the protocol and to attend required study training and visits
4. Male or female subjects
5. Age 18-75
6. Motor incomplete SCI
7. Level of lesion: T10 and above, based on AIS level, preservation of sacral function
8. Focal spinal cord disorder caused by either trauma or non-traumatic and non-progressive condition (like hemorrhage, benign tumor)
9. Minimum 3 months of recovery after SCI, maximum 2 years after trauma
10. Completed in-patient rehabilitation program
11. WISCI II, level >2 (0-20 items): assistance of one or more persons. Ability to walk at least 10 meters
12. Stable medical and physical condition.
13. Adequate care-giver support and access to appropriate medical care in patient's home community

Exclusion Criteria:

1. Enrollment of the investigator, his/her family members, employees and other dependent persons
2. Limitation of standing and walking function based on accompanying (CNS) disorders
3. Cardiovascular disorders restricting physical training or peripheral nerve disorders
4. Implanted technical devices (pacemaker, defibrillator)
5. History of significant autonomic dysreflexia
6. Cognitive disorders/brain damage
7. Drug refractory epilepsy
8. Severe joint contractures disabling or restricting lower limb movements
9. Haematological disorders with increased risk of bleeding during surgical interventions
10. Participation in another study with investigational drug within the 30 days preceding and during the present study
11. Congenital or acquired lower limb abnormalities (affection of joints and bone)
12. Women who are pregnant or breast feeding or planning a pregnancy during the course of the study
13. Lack of safe contraception
14. Inability of the participant to follow the procedures of the study, e.g. due to language problems, psychological problems, dementia etc.
15. Known or suspected non-compliance, drug or alcohol abuse
16. Current or prior malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in 6 Minute Walk Test at baseline and 6 months post intervention | preoperative, 6 months post intervention
  Standardized test. Patient is asked to walk for 6 minutes. Result is the distance covered

SECONDARY OUTCOMES:
Change in 10 Meter Walking Test towards baseline | preoperative, early postop, before discharge, 1,3,6 months follow-up
  Standardized test. Patient is asked to walk 10 meters as quickly as possible. Result is the speed (m/s)
Change in Timed Up and Go test (TUG) towards baseline | preoperative, early postop, before discharge, 1,3,6 months follow-up
  Standardized test. Patient is asked to stand up from a sitting into Standing Position and walk 3 m and return to seated position. Result ist time.
Kinematic assessment during overground and treadmill walking | preoperative, early postop, before discharge, 1,3,6 months follow-up
  Individuals are secured using the FLOAT.
Change in Spinal cord Independence measure (SCIM III) towards baseline | preoperative, early postop, before discharge, 1,3,6 months follow-up
  Standardized tool measuring the degree of independence of the subject. Result is score.
Change in Walking index for spinal cord injury (WISCI II) towards baseline | preoperative, early postop, before discharge, 1,3,6 months follow-up
  Standardized tool measuring the subject's ability to walk. Result is score.
Long-term monitoring of physical activity | Continuously between discharge and 6 months follow-up
  Wearable and wireless sensors are mounted to the patient and wheelchair for constant monitoring of physical activity
Electrophysiology | Baseline and several time-points throughout the study.
  SSEPs, MEPs, DBS-EPs, LFPs, EMG
Changes in Electroencephalography towards baseline | preoperative, intraoperative, early postop, 6 months follow-up
  Evaluation for the occuracne of EEG abnormalities
Change in Quality of life towards baseline | preoperative, 1,3,6 months follow-up
  Standardized QOL tool (SF-36). Result is score.
Change in lower urinary tract function towards baseline | preoperative, 6 months follow-up
  Standardized tools QUALIVEEN, bladder diary, urodynamic assessments, renal and bladder ultrasound.
Change in sexual functions towards baseline | preoperative, 1,3,6 months follow-up
  Use of the standardized tools FSFI (Female Sexual Function Index), result is score respectively IIEF (International Index of Erectile Function), result is score
Change in spasticity towards baseline | preoperative, early postop, before discharge, 1,3,6 months follow-up
  Use of the standardized tool MAS (Modified Ashword Scale). Result is score.
Changes in ASIA impairment scale (AIS) | preoperative, early postop, before discharge, 1,3,6 months follow-up
  Assment of neurological status of individual with SCI
Change in Upper limb Sensation, Strength and Prehension towards baseline | preoperative, 6 months follow-up
  Standardized tool GRASSP
Change in sleepiness towards baseline | preoperative, 1,3,6 months follow-up
  Standardized tool Epworth Sleepiness Scale
Change in Fatigue towards baseline | preoperative, 1,3,6 months follow-up
  Standardized tool Fatigue Severity Scale
Change in pain sensation towards baseline | preoperative, 1,3,6 months follow-up
  Standardized tools EPAF and SCIPI
Change in 6 Minute Walk Test at other timepoints towards baseline | Screening, early postop, before discharge, 1,3 months follow-up
  Standardized test. Patient is asked to walk for 6 minutes. Result is the distance

CONTACTS AND LOCATIONS:
Overall Officials: Lennart H Stieglitz, MD, Principal Investigator — University Hospital Zurich, Neurosurgery
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hofer AS, Stieglitz LH, Bolliger M, Filli L, Cathomen A, Willi R, Lerch I, Krusi I, Giagiozis M, Meyer C, Schubert M, Hubli M, Kessler TM, Demko L, Baumann CR, Imbach L, Oertel MF, Prusse A, Kiseleva A, Regli L, Schwab ME, Curt A. Cuneiform Nucleus Stimulation Can Assist Gait Training to Promote Locomotor Recovery in Individuals With Incomplete Tetraplegia. Ann Neurol. 2025 Sep 10. doi: 10.1002/ana.78026. Online ahead of print. PMID 40927915
- [Derived] Stieglitz LH, Hofer AS, Bolliger M, Oertel MF, Filli L, Willi R, Cathomen A, Meyer C, Schubert M, Hubli M, Kessler TM, Baumann CR, Imbach L, Krusi I, Prusse A, Schwab ME, Regli L, Curt A. Deep brain stimulation for locomotion in incomplete human spinal cord injury (DBS-SCI): protocol of a prospective one-armed multi-centre study. BMJ Open. 2021 Sep 30;11(9):e047670. doi: 10.1136/bmjopen-2020-047670. PMID 34593490